CLINICAL TRIAL: NCT04621721
Title: Home-Based Physical Activity Intervention for Taxane-Induced CIPN
Acronym: B-HAPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00040035; 1R01CA229681-01A1 (NIH)
Record Dates: First submitted 2020-08-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Female; Chemotherapy-induced Peripheral Neuropathy; Gait Disorders, Neurologic; Balance; Distorted; Muscle Weakness
MeSH Terms: conditions — Gait Disorders, Neurologic; Muscle Weakness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the investigator, co-investigators, statistician and data collectors will be blinded to study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention will consist of a 16-week, home-based gait/balance training and progressive resistance exercises for lower extremities using resistance power bands. Participants will be given the home-based gait/balance training and progressive resistance exercise training access via a link or by DVD, and the resistance training band, and wide, firm foam surface. The intervention group will begin with light warm-up and stretching activity then a 10 minute each of gait/balance and 10 minutes of resistive (strength) training components. The program begins with light stretching to address any range of motion limitations that may affect ability to maintain balance and postural stability, and consisted of hamstring quadricep, gastroc, and soleus stretches. During stretching exercises, participants held each stretch for 10-15 seconds, repeating each stretch 2-3 times for each lower extremity. Stretching exercises do not change during the intervention.
  Interventions: Behavioral: Gait/balance & resistive exercise
- Attention Control Group (Active Comparator): The Attention Control group will receive an educational intervention via a journal in which to record their clinic appointments, and standardized American Cancer Society pamphlets which have been adjusted to fit within the journal binding for easy reference. At each data collection encounter, the intervention research assistant will discuss the information in each pamphlet, allowing time for questions related to the material. The educational materials consist of 1) Emotions and Breast Cancer; 2) Body Image and Sexuality After Breast Cancer; 3) Follow up Care After Breast Cancer Treatment; 4) Nutrition and Cancer. Sessions last approximately 45-60 minutes and occur at the same intervals as the intervention group and will precede data collection. Attention Control group participants will receive telephone calls every other week which will entail a social visit and reminder of data collection/attention intervention appointments to further equalize contact.
  Interventions: Behavioral: Gait/balance & resistive exercise

INTERVENTIONS:
Behavioral: Gait/balance & resistive exercise — Walking forward and back, walking with head motion, static standing, Standing Partial Tandem, Tandem Standing heel to toe, Standing with head turns Single leg stance and March in place. Resistance exercises include: calf raises, lunges, supine leg curls and extensions.

SUMMARY:
This two-group, randomized control trial (RCT) will test the effects of a home-based, 16 week gait/balance training plus resistance (exercise bands) exercise program as compared to an educational cancer survivorship attention control condition to address persistent taxane-induced peripheral neuropathy in 312 patients treated for invasive breast cancer with taxanes at 1 year or more after completion of therapy. Assessments of lower extremity muscle strength, gait/balance, nerve conduction, neuropathy symptoms, and quality of life (QOL) will be performed.

The proposed exercise intervention addresses gait/balance impairments and motor (resistance) components of taxane-induced peripheral neuropathy. The mechanism by which the intervention achieves the proposed outcomes is though 1) increasing endoneurial blood flow to peripheral nerves and mitochondria resulting in reduction in neuropathic symptoms (including pain) and clinical manifestations of peripheral neuropathy, while improving gait/balance in those with persistent neuropathy; 2) The subsequent increase in nutrient supply allows the mitochondria to function more efficiently, and may alleviate the neuropathic manifestations of taxane-induced peripheral neuropathy. 15

This is the first study proposing to test the home-delivery of an exercise intervention specifically aimed at persistent (long-term) taxane-induced neuropathy. If successful, this study will provide the only evidence-based intervention for patients suffering from persistent neuropathy from neurotoxic chemotherapy. Additionally, the home-delivery format makes this intervention easily translated into clinical practice.

Specific Aims:

In a sample of patients who completed a taxane-containing chemotherapy regimen (> 1 year) for breast cancer and who have a persistent neuropathy (VAS score of > 3) the specific aims of this RCT are:

1. To test the efficacy of a 16-week -delivered program of gait/balance training plus resistance exercise, compared to an educational attention control condition in increasing muscle strength, improving gait/balance and nerve conduction parameters, decreasing the severity of taxane-induced peripheral neuropathy symptoms, and increasing quality of life.
2. To evaluate for differences in muscle strength, gait/balance, sensory (sural) and motor (peroneal) nerve conduction, peripheral neuropathy symptoms, and quality of life (QOL) between patients who receive the exercise program, compared to those in an educational attention control condition controlling for age, BMI, taxane cycles and intervals, neuropathic pain, neuropathy/pain medications, current resistance exercise participation and falls/near falls experienced.

DETAILED DESCRIPTION:
The use of taxanes in breast cancer chemotherapy regimens is considered standard first line therapy.1 However, taxanes are known to induce peripheral neuropathy, from 59-87% for paclitaxel and from 11-64% for docetaxel. 2-4 Sensory manifestations can include pain; numbness, tingling, & burning; diminished proprioception, and decreased vibration and touch sensation. 5-6 Motor symptoms such as lower extremity muscle weakness and impaired balance has been reported. 7 Currently, peripheral neuropathy remains a significant toxicity resulting in taxane chemotherapy dose reductions or discontinuation, with no evidence-based preventative or treatment strategies are available. 8 Taxanes induce sensory and motor neuropathy by inducing both mitochondrial and vascular dysfunction.9 In rodents, treatment with taxanes resulted in swollen, vacuolated axonal mitochondria that are functionally impaired, producing a chronic energy deficit.10 In addition, toxic effects to the endothelial cells of the vasa nervorum (small arterioles that supply peripheral nerves) in the dorsal root ganglia attenuates blood flow to neurons, resulting in endothelial cell death. 11 These findings suggest that both mitochondrial impairment and vascular damage are major mechanisms that underlie the development of taxane-induced peripheral neuropathy, manifesting as sensory manifestations and neuropathic pain. 9-12

Mitochondrial and vascular dysfunctions lead to sensory loss and reduced muscle strength, functions dependent upon cellular mitochondria to generate energy in the form of ATP (adenosine triphosphate). Thus, mitochondrial dysfunction results in the loss of energy-generating capability, and vascular impairment deprives muscle and nerve cells of oxygen-rich nutrients, further impairing neuronal function. A limited number of human and animal studies have demonstrated that exercise stimulates endothelium-dependent vasodilation and vascular endothelial growth factor (VEGF) expression, increasing endoneurial blood flow and energy generating capacity through mitochondrial protein synthesis and glycolysis, 13, 14

The proposed exercise intervention addresses gait/balance impairments and motor (resistance) components of taxane-induced peripheral neuropathy. The mechanism by which the intervention achieves the proposed outcomes is though 1) increasing endoneurial blood flow to peripheral nerves and mitochondria resulting in reduction in neuropathic symptoms (including pain) and clinical manifestations of peripheral neuropathy, while improving gait/balance in those with persistent neuropathy; 2) The subsequent increase in nutrient supply allows the mitochondria to function more efficiently, and may alleviate the neuropathic manifestations of taxane-induced peripheral neuropathy.

Specific Aims:

In a sample of patients who completed a taxane-containing chemotherapy regimen (> 1 year) for breast cancer and who have a persistent neuropathy (VAS score of > 3) the specific aims of this RCT are:

1. To test the efficacy of a 16-week -delivered program of gait/balance training plus resistance exercise, compared to an educational attention control condition in increasing muscle strength, improving gait/balance and nerve conduction parameters, decreasing the severity of taxane-induced peripheral neuropathy symptoms, and increasing quality of life.
2. To evaluate for differences in muscle strength, gait/balance, sensory (sural) and motor (peroneal) nerve conduction, peripheral neuropathy symptoms, and quality of life (QOL) between patients who receive the exercise program, compared to those in an educational attention control condition controlling for age, BMI, taxane cycles and intervals, neuropathic pain, neuropathy/pain medications, current resistance exercise participation and falls/near falls experienced

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivors (>21) with who completed treatment for invasive breast cancer with taxane-based chemotherapy, and who have a peripheral neuropathy score of > 3 by VAS rating consistent with studies of diabetic peripheral neuropathy.

Exclusion Criteria:

* any disease (e.g. diabetes, HIV) that results in peripheral neuropathy or muscle weakness (such as chronic fatigue syndrome, multiple sclerosis, spinal cord tumors or injuries, stroke,); any disease that would preclude exercise (preexisting cardiopulmonary disease, bone metastasis). Individuals with symptomatic lymphedema or advanced disease at high risk for bone metastases and pathologic fracture will be excluded.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer survivors age 21 and above
Enrollment: 312 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Gait Change | Change from Baseline to week 16
  Gait analysis will be performed using a GAITRite System with 3D motion capture with integrated force platform. Gait variables to be used in analysis are ankle plantar/flexor torque
Balance Change | Change from Baseline to week 16
  Balance analysis will be performed using the Neurocom Balance Master Sensory Organization Test
Change in Lower Extremity Muscle Strength | Change from Baseline to week 16
  Isokinetic dynamometry (Biodex 3.0) Hip flexors, hip abductors, knee flexors, knee extensors, and ankle dorsiflexors will be tested
Change in Lower Extremity Nerve Conduction | Change from Baseline to week 16
  Nerve conduction studies of the sural & peroneal nerve action potentials will be tested by Dr. Vu, USF Department of Neurology.
Change in Neuropathy Symptoms | Change over time from Baseline to 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  FACT-Taxane Additional Concerns subscale53 Addresses symptoms specific to neuropathy. Likert scale: 0 (not at all) - 4 (very much).
Neuropathy Quality of Life | Change over time from Baseline to 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  FACT-Taxane (version 4) 54 A total Quality of Life score can be obtained by summing the subscale scores and will be used for in the data analysis.

SECONDARY OUTCOMES:
Change in Neuropathic Pain | Change over time from Baseline to 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  Brief Pain Inventory assesses severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours
Change in Body Mass Index | Change from Baseline to week16
  A portable Tanita Body Composition Analyzer will be used to obtain each participant's weight and body mass index (BMI) through bioelectrical impedance.
Change in Neuropathy or Pain Medications | Change over time from Baseline to 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  Medications used for neuropathy pain will be monitored and documented throughout the study, and coded into drug classifications, and dosage change/no change tracked for analysis
Change in Falls or near falls in last month | Change over time from Baseline to 4 weeks, 8 weeks, 12 weeks, and 16 weeks
  participant will self-report (yes/no) if they have fallen or had a near fall within the last month.

OTHER OUTCOMES:
Participant age | Baseline
  participant will provide their age by self-report
Taxane cycles | Baseline
  Number of taxane cycles received and interval since last treatment will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozorio Dutra SV, Schwab L, Coury J, Ji M, Visovsky C. Process evaluation protocol plan for a home-based physical activity intervention versus educational intervention for persistent taxane-induced peripheral neuropathy (B-HAPI study): a randomized controlled trial. BMC Cancer. 2024 Jun 27;24(1):777. doi: 10.1186/s12885-024-12444-x. PMID 38937667
- [Derived] Teran-Wodzinski P, Haladay D, Vu T, Ji M, Coury J, Adams A, Schwab L, Visovsky C. Assessing gait, balance, and muscle strength among breast cancer survivors with chemotherapy-induced peripheral neuropathy (CIPN): study protocol for a randomized controlled clinical trial. Trials. 2022 Apr 27;23(1):363. doi: 10.1186/s13063-022-06294-w. PMID 35477489